CLINICAL TRIAL: NCT03847857
Title: A Multicenter Prospective Randomized Controlled Study of Porcine Fibrin Sealant in Preventing Cervical Anastomotic Leakage for Esophageal or Junctional Carcinoma. (PLACE030)
Brief Title: Study of Porcine Fibrin Sealant in Preventing Cervical Anastomotic Leakage (PLACE030)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yang Hong, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2019-011-01
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Anastomotic Leak
Keywords: Esophageal Cancer; Anastomotic Leak
MeSH Terms: conditions — Esophageal Neoplasms; Anastomotic Leak | interventions — Bioseal

STUDY DESIGN:
Intervention Model Description: A(Surgery+PFS) Arm A consists of the concurrent application of Porcine Fibrin Sealant (PFS) on the gastroesophageal anastomosis during Mckeown surgery . Biological/Vaccine: Porcine Fibrin Sealant (PFS) 2.5ml Porcine Fibrin Sealant will be instilled over the cervical anastomose line.
  B(Surgery)Arm B for conventional anastomosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery+PFS (Experimental): Arm A consists of the concurrent application of Porcine Fibrin Sealant (PFS) on the gastroesophageal anastomosis during McKeown esophagectomy.
  Interventions: Biological: Porcine Fibrin Sealant (PFS); Procedure: McKeown esophagectomy
- Surgery (Placebo Comparator): Arm B underwent conventional anastomosis during McKeown esophagectomy.
  Interventions: Procedure: McKeown esophagectomy

INTERVENTIONS:
Biological: Porcine Fibrin Sealant (PFS) — McKeown esophagectomy will be performed for patients with resectable thoracic esophageal carcinoma or gastroesophageal junction cancer. At last, 2.5ml Porcine Fibrin Sealant will be instilled over the cervical anastomose line.
  Other Names: Bioseal®
  Arms: Surgery+PFS
Procedure: McKeown esophagectomy — McKeown esophagectomy including open or minimally invasive esophagectomy will be performed for patients with resectable thoracic esophageal carcinoma or gastroesophageal junction cancer. Two-field lymphadenectomy with total mediastinal lymph node dissection is performed during surgery.

SUMMARY:
The primary objective is to evaluate the efficacy and assess the role of Porcine Fibrin Sealant (Bioseal®) in preventing cervical anastomotic leakage after esophagectomy in the patients with resectable thoracic esophageal cancer and gastroesophageal junction cancer.

DETAILED DESCRIPTION:
Esophageal cancer (EC) is the most common cancers in the world, with more than 16,910 new cases and 15,690 deaths annually worldwide. Every year in China, no matter new cases or deaths account for more than half of the world. Currently, surgery is the most important and effective treatment for esophageal cancer. According to the recommendation in Chinese Experts' Consensus on Esophageal Cancer Radical Surgery (year 2017), the rightapproach esophagectomy should be adopted, in order to achieve radical lymph nodes dissection and improve the surgical outcomes. So Mckeown procedure is recommended preferentially. However, esophageal resection for cancer has been associated perioperative mortality. One of the major perioperative complications that affect morbidity and mortality in these patients is esophageal anastomotic leakage. Moreover, it was reported that the leakage incidence of cervical anastomosis after esophageal cancer resection was significantly higher than that of intrathoracic anastomosis. Therefore, how to minimize the incidence of esophageal anastomotic leaks in esophagectomy is particularly important, especially for Mckeown surgery.

In recent years, the prognostic outcome of esophageal cancer has been improved due to advances in surgical technique. However, esophageal anastomotic leakage is still one of the most serious complications following esophagectomy, with an incidence around 5% to 40%. For example, a research based on Japanese national database showed that the rate of anastomotic leakage after esophagectomy was 13.3%. A recent phase 3 clinical trial, the ChemoRadiotherapy for Oesophageal Cancer Followed by Surgery Study (CROSS) reported an anastomotic leak rate of 26.1% after esophagectomy. Meanwhile, data from the investigator's center indicated that the leakage rate after esophagectomy was around 21.0%. Furthermore, anastomotic leakage following esophagectomy could seriously increase early mortality. According to the previous study, the risk of perioperative 90-day death was three times in patients with anastomotic leakage after esophagectomy than those without leaks (18.2% vs. 6.2%, P=0.003), and hospitalization was significantly increased.

Bioseal® (Guangzhou Bioseal Biotech Co., Ltd., China) is a porcine-derived fibrin sealant that has been widely used in various surgical procedures to assist in hemostasis for more than a decade. This type of fibrin sealant is made from biologically porcine-derived thrombin and fibrinogen, and is designed to form a stable fibrin clot by simulating the final pathway of the coagulation cascade. The fibrin clot will form a gel-like material on the surface of the surgical wound, which can not only directly block the tissue defect, but also promote the healing of the wound by using the fibrin network as the matrix where the fibroblasts and capillary endothelial cells can proliferate to form granulation. Therefore, Bioseal® have been reported to be used as sealing agent as well as wound healing agent during surgery in some studies.

In the recent years, some investigators have attempted to use the fibrin sealant to treat or prevent gastrointestinal leakage after enterectomy, gastrectomy, esophagectomy, or pancreaticoduodenectomy. The preliminary results show application of fibrin sealant may lower the chances of anastomotic leakage. Hence, it can diminish the mortality and morbidity of those patients with gastrointestinal reconstructions.

In 2004, a study conducted by Nguyen both in vitro and in vivo, found that application of fibrin sealant over gastric bypass could reduce the postoperative anastomotic leakage. Among the 16 animals (pigs) undergoing laparoscopic gastric bypass, 10 cases were applied with fibrin sealant on their primary anastomosis, and no anastomotic leakage or related complications was found. Five of the other 6 cases in control group had fistula or intra-abdominal abscess. Moreover#the follow-up study in humans showed that 66 patients in whom fibrin sealant was used as reinforcement on a primary anastomosis were all free of anastomotic leakage. In China, some studies also reported fibrin sealant could prevent anastomotic leakage for patients undergoing resection of rectal carcinoma or pancreato-biliary tumors.

As to esophagectomy, only few pilot studies have reported the similar attempts to prevent anastomotic leakage by using fibrin sealant. In 2007, Ling reported that application of fibrin sealant while implanting an esophageal stent under endoscopy was an effective approach for treating the postoperative esophageal anastomotic leakage. The studies conducted by Celal also showed that endoscopic treatment combined with fibrin sealant could be considered as a valuable option for the management of postoperative esophageal anastomotic leakage with a high degree of technical feasibility and safety. However, studies focusing on the role of fibrin sealant in the prevention of cervical leakage after esophagectomy are few.

In 2007, a prospective clinical trial conducted by Upadhyaya enrolled 45 infant patients who underwent esophagectomy for congenital esophageal atresia (EA) with tracheoesophageal fistula (TEF). In that study, a total of 52 patients were divided into two groups. In Group A, patients received fibrin sealant as reinforcement on a primary end-to-end esophageal anastomosis. In group B, fibrin glue was not used. In the final analysis, the overall rate of postoperative leakage is 26.9% (12/45), including 9.1% (2/22) in group A and 43% (10/23) in group B (p=0.017). In 2009, Saldaña-Cortés conducted a similar research but on puerile esophagectomy for caustic injury. Results showed that the postoperative cervical anastomotic dehiscence and leakage were observed in 28.5% of patients who received fibrin sealant in the study group and 50% of those in the control group. Both of those two studies indicated that fibrin glue, when used as a sealant for cervical esophageal anastomosis, could reduce the risk of leakage.

However, there is still no large-scale clinical trial investigating the use of fibrin sealant to prevent cervical anastomotic leakage after esophagectomy for esophageal cancer all over the world. The purpose of this study is to assess the role of fibrin glue (Bioseal®) in the prevention of leakage at the cervical esophageal anastomosis for esophageal cancer patients undergoing Mckeown surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of squamous cell carcinoma or adenocarcinoma of thoracic esophageal carcinoma or gastroesophageal junction cancer with Stage T1-4aN0-3M0, according to 8th edition of Union for International Cancer Control (UICC) staging system
2. More than 6 months of expected survival
3. Age ranges from 18 to75 years
4. Absolute white blood cells count ≥4.0×109/L, neutrophil ≥1.5×109/L, platelets ≥100.0×109/L, hemoglobin ≥90g/L, and normal functions of liver and kidney.
5. WHO performance status (PS) of 0-1
6. Informed consent will be obtained before the study

Exclusion Criteria:

1. Patients who have undergone definitive chemoradiotherapy
2. Patients with concomitant hemorrhagic disease
3. Patients with other uncontrollable status that cannot tolerate surgery
4. Patients with known hypersensitivity to the porcine fibrin sealant product
5. Pregnant or breast feeding
6. Patients cannot signed the informed consent document because of psychological quality, family and social factors
7. Patients with concomitant peripheral neuropathy, whose CTC status is 2 or even more
8. Have a history of diabetes over 10 years and with poorly controlled blood sugar level
9. Patients with serious cardiac, respiratory, hepatic, renal,hematologic, immunological disease or cachexy, who cannot tolerate surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative cervical anastomotic leakage | within the first 3 months after esophagectomy
  Incidence of postoperative cervical anastomotic leakage Cervical anastomotic leakage will be diagnosed based on a combination of clinical presentation, radiological findings, and/or endoscopic findings within the first 3 months after the operation.

SECONDARY OUTCOMES:
Overall survival Overall survival (OS) | At end of trial- up to 2 years in follow up
  Overall survival Overall survival (OS) is defined as the time period from the date of enrollment to the date of death or the last follow up
Disease Free Survival Disease-free survival (DFS) | At end of trial- up to 2 years in follow up
  Disease Free Survival Disease-free survival (DFS) is defined as the time period from the date of R0 resection to the date of disease recurrence or death.
Postoperative Complications | within the first 3 months after esophagectomy
  Postoperative complications will be recorded after each esophagectomy

CONTACTS AND LOCATIONS:
Overall Officials: Hong Yang, Ph.D.,M.D., Principal Investigator — Sun Yat-sen University Cancer Cente
Locations (6):
- China (6):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Jieyang Affiliated Hospital, Sun Yat-sen University, Jieyang, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Shantou, Guangdong
  - Zhongshan Peoples Hospital, Zhongshan, Guangdong
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Shanghai Chest Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Jones CE, Watson TJ. Anastomotic Leakage Following Esophagectomy. Thorac Surg Clin. 2015 Nov;25(4):449-59. doi: 10.1016/j.thorsurg.2015.07.004. Epub 2015 Sep 8. PMID 26515945
- [Background] Low DE. Diagnosis and management of anastomotic leaks after esophagectomy. J Gastrointest Surg. 2011 Aug;15(8):1319-22. doi: 10.1007/s11605-011-1511-0. Epub 2011 May 10. PMID 21557015
- [Background] Zhou C, Ma G, Li X, Li J, Yan Y, Liu P, He J, Ren Y. Is minimally invasive esophagectomy effective for preventing anastomotic leakages after esophagectomy for cancer? A systematic review and meta-analysis. World J Surg Oncol. 2015 Sep 4;13:269. doi: 10.1186/s12957-015-0661-z. PMID 26338060
- [Background] Law S, Fok M, Chu KM, Wong J. Comparison of hand-sewn and stapled esophagogastric anastomosis after esophageal resection for cancer: a prospective randomized controlled trial. Ann Surg. 1997 Aug;226(2):169-73. doi: 10.1097/00000658-199708000-00008. PMID 9296510
- [Background] Yuan Y, Zeng X, Hu Y, Xie T, Zhao Y. Omentoplasty for oesophagogastrostomy after oesophagectomy. Cochrane Database Syst Rev. 2014 Oct 2;2014(10):CD008446. doi: 10.1002/14651858.CD008446.pub3. PMID 25274134
- [Background] Takeuchi H, Miyata H, Gotoh M, Kitagawa Y, Baba H, Kimura W, Tomita N, Nakagoe T, Shimada M, Sugihara K, Mori M. A risk model for esophagectomy using data of 5354 patients included in a Japanese nationwide web-based database. Ann Surg. 2014 Aug;260(2):259-66. doi: 10.1097/SLA.0000000000000644. PMID 24743609
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Liu Q, Chen J, Wen J, Yang H, Hu Y, Luo K, Tan Z, Fu J. Comparison of right- and left-approach esophagectomy for elderly patients with operable thoracic esophageal squamous cell carcinoma: a propensity matched study. J Thorac Dis. 2017 Jul;9(7):1883-1890. doi: 10.21037/jtd.2017.06.22. PMID 28839986
- [Background] Rutegard M, Lagergren P, Rouvelas I, Lagergren J. Intrathoracic anastomotic leakage and mortality after esophageal cancer resection: a population-based study. Ann Surg Oncol. 2012 Jan;19(1):99-103. doi: 10.1245/s10434-011-1926-6. Epub 2011 Jul 19. PMID 21769467
- [Background] Ederle A, Scattolini C, Bulighin G, Benini L, Orlandi PG, Talamini G, Vantini I. Does the combination of a human fibrin sealant with ranitidine accelerate the healing of duodenal ulcer? Ital J Gastroenterol. 1991 Jul-Aug;23(6):354-6. PMID 1742526
- [Background] Nguyen NT, Nguyen CT, Stevens CM, Steward E, Paya M. The efficacy of fibrin sealant in prevention of anastomotic leak after laparoscopic gastric bypass. J Surg Res. 2004 Dec;122(2):218-24. doi: 10.1016/j.jss.2004.05.005. PMID 15555621
- [Background] Martin I, Au K. Does fibrin glue sealant decrease the rate of anastomotic leak after a pancreaticoduodenectomy? Results of a prospective randomized trial. HPB (Oxford). 2013 Aug;15(8):561-6. doi: 10.1111/hpb.12018. Epub 2012 Dec 27. PMID 23458447
- [Background] Tekinbas C, Erol MM, Akdogan R, Turkyilmaz S, Aslan M. Treatment of anastomotic leaks after esophagectomy with endoscopic hemoclips. J Thorac Cardiovasc Surg. 2009 Mar;137(3):766-7. doi: 10.1016/j.jtcvs.2008.01.052. Epub 2008 Sep 14. No abstract available. PMID 19258111
- [Background] Lee S, Ahn JY, Jung HY, Lee JH, Choi KS, Kim DH, Choi KD, Song HJ, Lee GH, Kim JH, Kim BS, Yook JH, Oh ST, Kim BS, Han S. Clinical outcomes of endoscopic and surgical management for postoperative upper gastrointestinal leakage. Surg Endosc. 2013 Nov;27(11):4232-40. doi: 10.1007/s00464-013-3028-y. Epub 2013 Jun 20. PMID 23783553
- [Background] Upadhyaya VD, Gopal SC, Gangopadhyaya AN, Gupta DK, Sharma S, Upadyaya A, Kumar V, Pandey A. Role of fibrin glue as a sealant to esophageal anastomosis in cases of congenital esophageal atresia with tracheoesophageal fistula. World J Surg. 2007 Dec;31(12):2412-5. doi: 10.1007/s00268-007-9244-7. PMID 17917772
- [Background] Saldana-Cortes JA, Larios-Arceo F, Prieto-Diaz-Chavez E, De Buen EP, Gonzalez-Mercado S, Alvarez-Villasenor AS, Prieto-Aldape MR, Fuentes-Orozco C, Gonzalez-Ojeda A. Role of fibrin glue in the prevention of cervical leakage and strictures after esophageal reconstruction of caustic injury. World J Surg. 2009 May;33(5):986-93. doi: 10.1007/s00268-009-9949-x. PMID 19234736